CLINICAL TRIAL: NCT04507074
Title: The Effect of Traction Forces on Changes in Biochemical Markers of Degeneration and Functional Parameters of the Spine in People With Obesity Suffering From Chronic Low Back Pain
Brief Title: The Effect of Traction Forces in People With Obesity Suffering From Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Principal Investigator, Marzena Ratajczak, assistant professor, Poznan University of Physical Education
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PoznanUPhyEd no. 3
Record Dates: First submitted 2020-07-06; First posted 2020-08-10 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Low Back Pain; Obesity
Keywords: biomarkers of low back pain; inflammation; disk degeneration; traction therapy; lumbar traction
MeSH Terms: conditions — Low Back Pain; Obesity; Inflammation; Intervertebral Disc Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients With Obesity (Experimental): 40 subjects aged 35-60 with simple obesity (BMI ≥ 30 kg / m2) and chronic low back pain.
  Interventions: Device: lumbar traction therapy
- Normal-Weight Patients (Active Comparator): 20 subjects aged 35-60 with normal body weight (BMI ≤ 24.9 and ≥ 18.5 kg/m2) suffering from chronic low back pain.
  Interventions: Device: lumbar traction therapy

INTERVENTIONS:
Device: lumbar traction therapy — The application of traction forces on the traction table (ST6567P-SEERSMEDICAL) will last 30 minutes a day for 4 weeks (continuous traction mode with a maximum strength of 30% of the patient's body weight).
  Other Names: lumbar traction

SUMMARY:
The purpose of the research study is to assess the impact of traction forces on changes in systemic markers concentrations of spinal structure damage in people with obesity. The research group will include 40 subjects aged 35-60 with simple obesity (BMI ≥ 30 kg / m2) and chronic lumbar spine pain syndrome.

The control group will consist of 20 subjects with normal body weight suffering from the same pain, at a similar age to the patients in the study group. Persons will be qualified for examination by a specialist in internal medicine and a physiotherapist.

To assess the degree of structural damage within the intervertebral disc and adjacent anatomical structures, patients will undergo magnetic resonance imaging of the lumbosacral spine (MRI 1.5T, standard in 3 projections). Patients will undergo traction therapy under the supervision of a physiotherapist. The application of traction forces on the traction table (ST6567P-SEERSMEDICAL) will last 30 minutes a day for 4 weeks (continuous traction mode with a maximum strength of 30% of the patient's body weight).

Twice, before and after therapy, the following will be assessed: (1) body composition (by DXA method), (2) other anthropometric indicators, (3) functional parameters of the spine: mobility (electrogoniometer), muscle bioelectric signal amplitude (electromyograph), soft tissue biophysical parameters (myotonometer), (4) pain threshold and intensity in the lumbar region (using an algometer and validated questionnaires), (5) disability caused by pain in the spine (Oswestry questionnaire), (6) blood biochemical indicators selected on the basis of the latest research on biomarkers of spinal damage (for this purpose, 25ml venous blood will be taken from the subjects).

Blood levels of interleukin-17, interleukin-4, interleukin-2 (IL-2), interleukin-10 (IL-10), differentiating growth factor 15 (GDF-15), leptin, adipsin, chemokine CCL5 (RANTES), stem cell growth factor β (SCGF-β), vascular endothelial growth factor (VEGF), neuropeptide Y, and chondroitin sulfate CS846 will be determined in the blood of the subjects. It is planned to assess the relationship of the studied biomarkers with the degree of disk degeneration, obesity, lean and fat body mass, pain intensity, and functional indicators of the spine. Patients will be asked to stop taking anti-inflammatory drugs during therapy and at least 24 hours prior to blood sampling.

DETAILED DESCRIPTION:
People suffering from obesity are particularly vulnerable to mechanical compression of the intervertebral discs, and as a result their degeneration, hernia and pressure on the nerve roots, which together cause inflammation and pain in the damaged area. This is a significant public health problem due to the 100% incidence of pain syndrome among people with obesity. The use of traction forces has beneficial effects on degenerated intervertebral discs, but there are no studies assessing the effectiveness of the traction method in relation to a group of obese people with back pain syndrome.

Beneficial biochemical changes in the blood, alleviation of pain, improvement of functional parameters of the spine are expected after application of traction forces to the patients in the mechanism of decompression of the destroyed and being in chronic inflammation intervertebral discs. Identification of biomarkers enabling to monitor the effects of therapies in patients with chronic back pain can become a contribution to change standards in the diagnosis of back pain and reorientation in its treatment to real causes.

ELIGIBILITY:
Inclusion Criteria:

1. Written consent to participate in the study,
2. Age: 35 - 60 years,
3. Obesity (BMI ≥ 30 kg / m2) or normal weight (BMI 18,5-29,9 kg/m2),
4. Stable body weight in the last month ± 2 kg,
5. Chronic low back pain.

Exclusion Criteria:

1. Secondary form of obesity;
2. Serious neurological defects (including large muscle losses, sensory disturbances in a large area of the lower limb, occurrence of cauda equina syndrome);
3. Surgery, post-accident mechanical injuries, history of spine fractures;
4. History of rheumatic disease (RA, ankylosing spondylitis, systemic lupus);
5. Osteoporosis;
6. Pain located in a location other than the spine which is more severe than the low back pain;
7. Poorly controlled type 2 diabetes;
8. Poorly controlled hypertension (mean systolic blood pressure> 140mmHg and / or average diastolic blood pressure> 90mmHg) during the last month and / or the necessity of modification of pharmacological treatment;
9. Lipid disorders requiring the introduction of pharmacological treatment in the last 3 months before observation or during observation;
10. Acute coronary event, unstable angina, stroke or transient cerebral ischemia in the last 6 months;
11. Features of heart failure in physical examination and / or additional tests (chest X-ray, echocardiography);
12. Clinically significant arrhythmias, conduction disorders, pacemaker implantation;
13. Fainting in an interview,
14. Chronic kidney disease with creatinine clearance <60mL / min / 1.73m2;
15. Clinically significant liver dysfunction (transaminases exceeding 3 times the normal range);
16. Acute or chronic, clinically apparent inflammatory process of the respiratory tract, inflammatory processes of the genitourinary system, inflammatory process in the head and neck;
17. Acute infection in the last month;
18. Cancer;
19. Alcohol abuse, drug addiction;
20. Pregnancy;
21. Uncontrolled mental illness that may falsify test results;
22. Other conditions which may pose any risk to the patient during the observation.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Interleukin-2, interleukin-4, interleukin-10, interleukin-17, RANTES, differentiating growth factor 15 (GDF-15) [pg/ml] | pre-intervention
  ELISA
Interleukin-2, interleukin-4, interleukin-10, interleukin-17, RANTES, differentiating growth factor 15 (GDF-15) [pg/ml] | 48 hours after the intervention
  ELISA
Stem cell growth factor β [ng/ml] | pre-intervention
  ELISA
Stem cell growth factor β [ng/ml] | 48 hours after the intervention
  ELISA
Leptin [ng/ml] | pre-intervention
  ELISA
Leptin [ng/ml] | 48 hours after the intervention
  ELISA
Adipsin [pg/ml] | pre-intervention
  ELISA
Adipsin [pg/ml] | 48 hours after the intervention
  ELISA
Neuropeptide Y [pg/ml] | pre-intervention
  ELISA
Neuropeptide Y [pg/ml] | 48 hours after the intervention
  ELISA
Vascular Endothelial Growth Factor [pg/ml] | pre-intervention
  ELISA
Vascular Endothelial Growth Factor [pg/ml] | 48 hours after the intervention
  ELISA
Chondroitin sulfate CS846 [ng/mL] | pre-intervention
  ELISA
Chondroitin sulfate CS846 [ng/mL] | 48 hours after the intervention
  ELISA

SECONDARY OUTCOMES:
Magnetic resonance imaging of the lumbosacral spine | pre-intervention
  MRI 1.5T
Total body fat content [%] | pre-intervention
  dual energy X-ray absorptiometry (DXA)
Total body fat content [%] | 48 hours after the intervention
  dual energy X-ray absorptiometry (DXA)
Lean body mass [kg] | pre-intervention
  dual energy X-ray absorptiometry (DXA)
Lean body mass [kg] | 48 hours after the intervention
  dual energy X-ray absorptiometry (DXA)
Mobility of the spine | pre-intervention
  electrogoniometer
Mobility of the spine | 48 hours after the intervention
  electrogoniometer
Muscle bioelectric signal amplitude | pre-intervention
  electromyograph
Muscle bioelectric signal amplitude | 48 hours after the intervention
  electromyograph
State of tension of erector spinae muscles [Hz] | pre-intervention
  Natural oscillation frequency [Hz], characterizing Tone or Tension will be assessed with myotonometer device.
Dynamic stiffness of erector spinae muscles [N/m] | pre-intervention
  Biomechanical properties will be assessed with myotonometer device.
Logarithmic decrement of natural oscillation, characterizing elasticity of erector spinae muscles | pre-intervention
  Biomechanical properties will be assessed with myotonometer device.
State of tension of erector spinae muscles [Hz] | 48 hours after the intervention
  Natural oscillation frequency [Hz], characterizing Tone or Tension will be assessed with myotonometer device.
Dynamic stiffness of erector spinae muscles [N/m] | 48 hours after the intervention
  Biomechanical properties will be assessed with myotonometer device.
Logarithmic decrement of natural oscillation, characterizing elasticity of erector spinae muscles | 48 hours after the intervention
  Biomechanical properties will be assessed with myotonometer device.
Pain threshold | pre-intervention
  algometer
Pain threshold | 48 hours after the intervention
  algometer
Pain intensity: questionnaire | pre-intervention
  visual analogue scale (VAS) pain intensity questionare (reporting a score on a 10-point scale, the minimum (0) means no pain and the maximum (10) means a worst pain imaginable
Pain intensity: questionnaire | 48 hours after the intervention
  visual analogue scale (VAS) pain intensity questionare (reporting a score on a 10-point scale, the minimum (0) means no pain and the maximum (10) means a worst pain imaginable
Disability caused by pain in the spine | pre-intervention
  Oswestry questionnaire. When completing the questionnaire, the subject answers questions concerning: pain intensity, independence, lifting objects, walking, sitting, standing, sleeping, social life, sexual activity and traveling. The answers to the questions help to classify how limited the functioning of the patient is while performing certain activities. Responses are graded from 0 to 5. The overall score is given on a 0-50 point scale, where the higher the score, the greater the disability.
Disability caused by pain in the spine | 48 hours after the intervention
  Oswestry questionnaire. When completing the questionnaire, the subject answers questions concerning: pain intensity, independence, lifting objects, walking, sitting, standing, sleeping, social life, sexual activity and traveling. The answers to the questions help to classify how limited the functioning of the patient is while performing certain activities. Responses are graded from 0 to 5. The overall score is given on a 0-50 point scale, where the higher the score, the greater the disability.

CONTACTS AND LOCATIONS:
Overall Officials: Marzena Ratajczak, PhD, Principal Investigator — Poznan University of Physical Education; Małgorzata Waszak, PhD, Study Chair — Poznan University of Physical Education
Locations (1):
- Poznan University of Physical Education, Poznan, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chow DHK, Yuen EMK, Xiao L, Leung MCP. Mechanical effects of traction on lumbar intervertebral discs: A magnetic resonance imaging study. Musculoskelet Sci Pract. 2017 Jun;29:78-83. doi: 10.1016/j.msksp.2017.03.007. Epub 2017 Mar 20. PMID 28347933
- [Background] Omarker K, Myers RR. Pathogenesis of sciatic pain: role of herniated nucleus pulposus and deformation of spinal nerve root and dorsal root ganglion. Pain. 1998 Nov;78(2):99-105. doi: 10.1016/S0304-3959(98)00119-5. PMID 9839819
- [Background] Maciaszek J, Skrypnik D, Ratajczak M, Stemplewski R, Osiński W, Bogdański P, Mądry E, Walkowiak J, Karolkiewicz J. Two aerobic exercise programs in management of back pain among middle-aged obese women: A randomized controlled study. Human Movement. 2016; 17(2): 72-79.
- [Background] Weber KT, Satoh S, Alipui DO, Virojanapa J, Levine M, Sison C, Quraishi S, Bloom O, Chahine NO. Exploratory study for identifying systemic biomarkers that correlate with pain response in patients with intervertebral disc disorders. Immunol Res. 2015 Dec;63(1-3):170-80. doi: 10.1007/s12026-015-8709-2. PMID 26440592
- [Background] Tarabeih N, Shalata A, Trofimov S, Kalinkovich A, Livshits G. Growth and differentiation factor 15 is a biomarker for low back pain-associated disability. Cytokine. 2019 May;117:8-14. doi: 10.1016/j.cyto.2019.01.011. Epub 2019 Feb 15. PMID 30776685
- [Background] Sowa GA, Perera S, Bechara B, Agarwal V, Boardman J, Huang W, Camacho-Soto A, Vo N, Kang J, Weiner D. Associations between serum biomarkers and pain and pain-related function in older adults with low back pain: a pilot study. J Am Geriatr Soc. 2014 Nov;62(11):2047-55. doi: 10.1111/jgs.13102. Epub 2014 Nov 3. PMID 25367206
- [Derived] Ratajczak M, Wendt M, Sliwicka E, Skrypnik D, Zielinski J, Kusy K, Krutki P, Waszak M. Subjective assessment and biochemical evaluation of traction therapy in women with chronic low back pain: does body mass index matter? A clinical study. BMC Musculoskelet Disord. 2023 Mar 16;24(1):196. doi: 10.1186/s12891-023-06300-5. PMID 36927409